CLINICAL TRIAL: NCT03876769
Title: A Phase II Trial of Tisagenlecleucel in First-line High-risk (HR) Pediatric and Young Adult Patients With B-cell Acute Lymphoblastic Leukemia (B-ALL) Who Are Minimal Residual Disease (MRD) Positive at the End of Consolidation (EOC) Therapy
Brief Title: Study of Efficacy and Safety of Tisagenlecleucel in HR B-ALL EOC MRD Positive Patients
Acronym: CASSIOPEIA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019G2201J; 2017-002116-14 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2019-03-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia
Keywords: CTL019; Kymriah; B-Cell Acute Lymphoblastic Leukemia; ALL; tisagenlecleucel; HR B-ALL EOC MRD; Minimal Residual Disease (MRD); Positive at the End of Consolidation (EOC)
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose of CTL019 (Experimental): Based on the subject's weight one of two possible dose ranges will be prepared for the subject:
  Subjects ≤ 50 kg: 0.2 to 5.0 x 10(6) CAR-positive viable T cells per kg body weight
  OR
  Subjects > 50 kg: 0.1 to 2.5 x 10(8) CAR-positive viable T cells
  Interventions: Biological: CTL019

INTERVENTIONS:
Biological: CTL019 — Based on the subject's weight, one of two possible dose ranges will be prepared for the subject:
  Subjects ≤ 50 kg: 0.2 to 5.0 x 10(6) CAR-positive viable T cells per kg body weight
  OR
  Subjects > 50 kg: 0.1 to 2.5 x 10(8) CAR-positive viable T cells

SUMMARY:
This is a single arm, open-label, multi-center, phase II study to determine the efficacy and safety of tisagenlecleucel in de novo HR pediatric and young adult B-ALL patients who received first-line treatment and are EOC MRD positive. The study will have the following sequential phases: screening, pre-treatment, treatment & follow-up, and survival. After tisagenlecleucel infusion, patient will have assessments performed more frequently in the first month and then at Day 29, then every 3 months for the first year, every 6 months for the second year, then yearly until the end of the study. Efficacy and safety will be assessed at study visits and as clinically indicated throughout the study. The study is expected to end in approximately 8 years after first patient first treatment (FPFT). A post-study long term follow-up safety will continue under a separate protocol per health authority guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. CD19 expressing B-cell Acute Lymphoblastic Leukemia
2. De novo NCI HR B-ALL who received first-line treatment and are MRD ≥ 0.01% at EOC. EOC bone marrow MRD will be collected prior to screening and will be assessed by multi-parameter flow cytometry using central laboratory analysis.
3. Age 1 to 25 years at the time of screening
4. Lansky (age < 16 years) or Karnofsky (age ≥ 16 years) performance status ≥ 60%
5. Adequate organ function during the screening period:

   A. Renal function based on age/gender B. ALT ≤ 5 times ULN for age C. AST ≤ 5 times ULN for age D. Total bilirubin < 2 mg/dL (for Gilbert's Syndrome subjects total bilirubin < 4 mg/dL)

   E. Adequate pulmonary function defined as:
   * no or mild dyspnea (≤ Grade 1)
   * oxygen saturation of > 90% on room air F. Adequate cardiac function defined as LVSF ≥ 28% confirmed by echocardiogram or LVEF ≥ 45% confirmed by echocardiogram or MUGA within 6 weeks of screening
6. Prior induction and consolidation chemotherapy allowed: 1st line subjects: ≤ 3 blocks of standard chemotherapy for first-line B-ALL, defined as 4-drug induction, Berlin-Frankfurt-Münster (BFM) consolidation or Phase 1b, and interim maintenance with high-dose methotrexate.

Exclusion Criteria:

1. M3 marrow at the completion of 1st line induction therapy
2. M2 or M3 marrow or persistent extramedullary disease at the completion of first-line consolidation therapy or evidence of disease progression in the peripheral blood or new extramedullary disease prior to enrollment. Patients with previous CNS disease are eligible if there is no active CNS involvement of leukemia at the time of screening.
3. Philadelphia chromosome positive ALL
4. Hypodiploid: less than 44 chromosomes and/or DNA index < 0.81, or other clear evidence of a hypodiploid clone
5. Prior tyrosine kinase inhibitor therapy
6. Subjects with concomitant genetic syndromes associated with bone marrow failure states: such as subjects with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Subjects with Down syndrome will not be excluded.
7. Subjects with Burkitt's lymphoma/leukemia (i.e. subjects with mature B-ALL, leukemia with B-cell [sIg positive and kappa or lambda restricted positivity] ALL, with FAB L3 morphology and /or a MYC translocation)
8. Has had treatment with any prior anti-CD19 therapy 9. Treatment with any prior gene or engineered T cell therapy

Other protocol-defined inclusion/exclusion may apply.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2027-10-19 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) rate without censoring for new anticancer therapy, including Stem Cell Transplantation (SCT) while in remission | 5 years after tisagenlecleucel infusion
  DFS is defined as the time from the date of tisagenlecleucel infusion to the date of the first documented morphological relapse, occurrence of secondary malignancy or death due to any cause.
Overall Survival (OS) rate | 4 years after tisagenlecleucel
  OS is defined as the time from date of first tisagenlecleucel infusion to the date of death due to any reason.

SECONDARY OUTCOMES:
Percentage of participants who are disease free without allogeneic stem cell transplant (SCT) | 12 months after last infusion
  Minimal Residual Disease (MRD) negative remission (complete remission (CR) or Complete remission with incomplete blood count recovery CRi)) at Month 12 without SCT after tisagenlecleucel infusion.
DFS rate with censoring for new anticancer therapy, including SCT, while in remission | 5 years
  Assessing the effect of tisagenlecleucel on DFS if new anticancer therapy is not available.
Percentage of participants achieving MRD negative CR or CRi at Month 3 | 3 months after the tisagenlecleucel infusion.
  Assessing the percentage of participants who achieved MRD negative complete response (CR) or Complete remission with incomplete blood count recovery (CRi) status as determined by central laboratory using multi-parameter flow cytometry.
Pediatric Quality of Life (PedsQL) | 5 years
  Patient reported outcome to assess quality of life in patients aged 8 and above. The 23 items PedQL (Pediatrics Quality of Life Inventory) measure core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning.
  Items measured include 1) Physical Functioning (8 items), 2) Emotional Functioning (5 items), 3) Social Functioning (5 items), and 4) School Functioning (5 items).
  Each item is measured on a 5 point Likert scale with 0 indicating "never" and 4 indicating "almost always".
  The Likert scores are reversed scored and linearly transform to a 0-100 scale with 0=100, 1-75, 2=50, 5=25, and 4=0. A higher score indicates better health-related quality of life (HRQoL).
European Quality of Life 5 dimensions (EQ-5D-3L & EQ-5D-Y)) | 5 years
  Patient reported outcome to assess health status in patients aged 8 and above. The EQ-5D (European Quality of Life -5 Dimensions) measures a wide range of health conditions and treatments; it is composed of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and a visual analogue scale (EQ-visual analogue scale [EQ-VAS]) that records the patient's self-rated overall health state.
  Respondents rate each of these 5 dimensions from "no problem", "some problem," or "extreme problem".
  The EQ-VAS records the respondents' self-related health on a vertical, visual analogue scale. The range for EQ-VAS is from 0 (=the worst health you can imagine) to 100 (=the best health you can imagine).
Impact of tisagenlecleucel on cognitive functioning using Computerized neurocognitive assessment: Detection test | 5 years
  Speed of performance (mean of the log10 transformed reaction times for correct responses)
Impact of tisagenlecleucel on cognitive functioning usingComputerized neurocognitive assessment: Identification test | 5 years
  This test measures the speed of performance (mean of the log10 transformed reaction times for correct responses)
Impact of tisagenlecleucel on cognitive functioning using Computerized neurocognitive assessment: Groton Maze Learning test | 5 years
  This test looks at the total number of errors made in attempting to learn the hidden pathways during a single session.
Impact of tisagenlecleucel on cognitive functioning using Computerized neurocognitive assessment: One Back test | 5 years
  This test measures the accuracy of performance (arcsine transformation of the square root of the percentage of correct responses). The test also measures the speed of performance (mean of the log10 transformed reaction times for correct responses).
Impact of tisagenlecleucel on cognitive functioning usingComputerized neurocognitive assessment: One card learning test | 5 years
  This test measures the accuracy of performance (arcsine transformation of the square root of the proportion of correct responses).
Percentage of participants with pre-existing antibodies | 8 years
  Prevalence of immunogenicity
Percentage of participants with anti-m CAR19 antibodies post infusion with tisagenlecleucel and % of patients without measureable anti-mCAR19 antibodies | 8 years
  Incidence of immunogenicity
Percentage of patients that have measureable anti-mCAR19 antibodies above patient specific cut-point (reported as a %) pre and post tisagenlecleucel infusion categorized by Day 28 response | 8 years
  Impact of immunogenicity on clinical response
tisagenlecleucel transgene concentration | 8 years
  Transgene concentration as detected by qPCR in target tissue
Expression of tisagenlecleucel | 8 years
  Summary of tisagenlecleucel CAR-positive viable T cells measured by flow cytometry in target tissue
Persistence of CAR (reported as copies/ug) categorized by the time to B-cell recovery (recovery < 3 months, >3 months to < 6months, > 6 months) | 8 years
  Relationship between B-cell recovery and transgene levels
Cmax; cellular kinetic parameter of tisagenlecleucel | 8 years
  The maximum (peak) observed in peripheral blood or other body fluid drug concentration after single dose administration (% or copies/μg)
Tmax; cellular kinetic parameter of tisagenlecleucel | 8 years
  The time to reach maximum (peak) peripheral blood or other body fluid drug concentration after single dose administration (days)
AUC0-29d and 84d; cellular kinetic parameter of tisagenlecleucel | 8 years
  The AUC from time zero to day 29 and 84 or other disease assessment days, in peripheral blood (% or copies/μg x days )
AUC0-Tmax; cellular kinetic parameter of tisagenlecleucel | 8 years
  The AUC from time zero to Tmax in peripheral blood (% or copies/μg x days)
T1/2; cellular kinetic parameter of tisagenlecleucel | 8 years
  The half-life associated with the elimination phase slope of a semi logarithmic concentration-time curve (days) in peripheral blood
Clast; cellular kinetic parameter of tisagenlecleucel | 8 years
  The last observed quantifiable concentration in peripheral blood (% or copies/μg)
Tlast; cellular kinetic parameter of tisagenlecleucel | 8 years
  The time of last observed quantifiable concentration in peripheral blood (days)
Impact of tisagenlecleucel dose on day 29 response | 8 years
  Clinical response summarized by quartile of administered doses
AUC 0 - 29d; cellular kinetic parameter of tisagenlecleucel | Day 29
  Impact of tisagenlecleucel exposure on day 29 response; The AUC from time zero to day 29 in peripheral blood (% or copies/μg x days )
Cmax: cellular kinetic parameter of tisagenlecleucel | Day 29
  Impact of tisagenlecleucel exposure on day 29 response; The maximum (peak) observed in peripheral blood or other body fluid drug concentration after single dose administration (% or copies/μg)
Tmax: cellular kinetic parameter of tisagenlecleucel | Day 29
  Impact of tisagenlecleucel exposure on day 29 response; The time to reach maximum (peak) peripheral blood or other body fluid drug concentration after single dose administration (days)
T1/2: cellular kinetic parameter of tisagenlecleucel | Day 29
  Impact of tisagenlecleucel exposure on day 29 response; The half-life associated with the elimination phase slope of a semi logarithmic concentration-time curve (days) in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (31):
  - Children s Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - City of Hope National Medical, Duarte, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Mattel Childrens Hospital UCLA, Los Angeles, California
  - Childrens Hospital of Orange County, Orange, California
  - Rady Children s Hospital, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Johns Hopkins All Childrens, St. Petersburg, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - James Whitcomb Riley Hospital For Children, Indianapolis, Indiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children s Mercy Hospital, Kansas City, Missouri
  - Hackensack Uni Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Childrens Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Univ of Texas Southwest Med Center, Dallas, Texas
  - Texas Children's Cancer and Hematology Center, Houston, Texas
  - Methodist Childrens Hospital, San Antonio, Texas
  - University of Utah Clinical Trials Office, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics Pharmacy/Drug Shipping Address, Madison, Wisconsin
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Novartis Investigative Site, Ghent, Belgium
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Roma, RM, Italy
- Netherlands (2):
  - Prinses Maxima Centrum voor Kinderoncologie, Utrecht, CS
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Esplugues, Barcelona, Spain
- Novartis Investigative Site, Gothenburg, Sweden
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Seftel MD. Hyper-CVAD: a regimen for all seasons. Lancet Haematol. 2020 Jul;7(7):e501-e502. doi: 10.1016/S2352-3026(20)30179-4. No abstract available. PMID 32589970